CLINICAL TRIAL: NCT04197089
Title: Pilot Study of the Biological Effects of Vitamin D in Patients With Resectable Urinary Tract Urothelial Carcinoma
Brief Title: Biological Effect of Vitamin D in Patients With Urothelial Carcinoma
Acronym: VitDURO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Centro Nacional de Investigaciones Oncologicas CARLOS III (Other); Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VitDURO-AECC17-01
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Urothelial Carcinoma
Keywords: Cancer; Urinary tract; Cystectomy; Vitamin D; Tissue phenotype
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Treatment stratified with 10.000 IU or 50.000 IU Vitamin D depending of baseline 25(OH)Vitamin D plasmatic levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D treatment (Experimental): Treatment with 10.000 IU or 50.000 IU Vitamin D weekly during 4 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — First dose of 10.000 IU Vitamin D at baseline visit for all patients; stratification of treatment (10.000 or 50.000 IU Vitamin D) depending base 25(OH)Vitamin D levels. Treatment weekly during 4 weeks before scheduled cystectomy
  Other Names: Cholecalciferol; Colecalciferol

SUMMARY:
The study population will be 50 women or men diagnosed with urothelial cancer candidates to undergo cystectomy as part of their antitumor treatment. The main objective of the study is to determine the biological effect of Vitamin D on tumor tissue phenotype; for thus, all subjects enrolled in the study will take Vitamin D supplementation 4 weeks prior undergoing surgery. Urothelial tissue will be obtained from the surgical procedure and will be studied for the Vitamin D effect on cancer cell, compared with that urothelial tissue biopsy obtained in the moment of cancer diagnosis.

DETAILED DESCRIPTION:
The study will enroll 50 patients (older than 18 and younger than 80 years old), recently diagnosed with urothelial cancer and candidates to undergo radical cystectomy or nephroureterectomy.

At the baseline visit, a blood sample will be obtained for 25OH-VitD analysis and all subjects will receive first dose of 10.000 IU Vitamin D. Depending of basal plasmatic Vitamin D value, patients will be stratified in either 10.000 IU treatment (25OH-VitD ≥ 20 ng/ml) or either 50.000 UI treatment dose (25OH-VitD < 20 ng/ml). Treatment will consist of 4 doses taken weekly before their scheduled cystectomy. Last study follow-up visit will be 4 weeks post-surgery. Urothelial tumor tissue collected on surgery will be used to evaluate the expression of tumor differentiation and Vitamin D markers, using genomics and proteomics approaches. Blood sample will also be collect throughout the study to evaluate the pharmacokinetics of Vitamin D in plasma and the expression of Vitamin D target genes in peripheral blood leukocytes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years
* Patients willing and able to read and understand the patient's information sheet and give their consent
* Histologically confirmed diagnosis of urothelial non-muscle-invasive bladder cancer (T1 high grade and/or carcinoma in situ), and patients with muscle-invasive or high urinary tract carcinoma without evidence of distant metastasis (T2-4N0M0)
* Candidate patients to undergo treatment by radical cystectomy or nephroureterectomy as part of conventional tumor treatment.
* Not having received any antitumor treatment during the 4 weeks prior the administration of Vitamin D
* Life expectancy longer than 6 months
* Karnofsky Index > 70%
* Confirmed adequate bone marrow, kidney and liver functions by:

  1. Leukocyte count > 4.000
  2. Platelet count > 100.000
  3. Haemoglobin levels > 10 gr/dl
  4. Serum bilirubin levels < 1,5X the upper limit of normality
  5. AST and ALT levels < 2,5X the upper limit of normality
  6. Alkaline Phosphatase levels < 5X the upper limit of normality
  7. Serum creatinine levels ≤ 2 mg/dl, and/or GFR ≥ ml/min/1.73m2 estimated by MDRD-4 IDMS or CKD-EPI evaluation
* Plasma calcium levels between 8.8 and 10.6 mg/dl, and 24 hours urine calcium levels between 100 and 300 mg/24h
* Women of childbearing potential should use a highly effective contraceptive method according the Clinical Trial Facilitation Group (such as combined hormonal contraceptives or IUD), and should continue its use for 90 days after the last dose of Vitamin D
* Males in fertile age, with potentially fertile partner, should use a contraceptive method such as sexual abstinence or barrier method (condom), throughout the clinical trial and up to 90 days after the end of treatment, or be vasectomized

Exclusion Criteria:

* Ade older than 80 years
* Patients with non-urothelial histology. Those with mixed histology may be included if the urothelial component is the predominant (> 50%)
* Administration of neoadjuvant chemotherapy
* Administration of radiotherapy during the period between TUR and surgery
* Medical history of another neoplasm diagnosed in the previous 3 years (except carcinoma in situ or non-melanoma cutaneous carcinoma). It may be included those patients with history of other neoplasms, provided that after receiving radical treatment do not relapsed
* History of hypersensitivity to Vitamin D
* History of renal lithiasis larger than 5 mm or symptomatic in the year prior its inclusion in the study, and/or nephrocalcinosis
* History of hypercalcemia and/or hypercalciuria
* Situation of hypervitaminosis (25-OH Vitamin D > 50 ng/ml)
* Previous treatment with Vitamin D in the last 6 months
* Chronic treatment with corticosteroids
* Other serious diseases or medical processes such as: infection that requires systemic anti-infective treatment or not controlled serious medical processes, including severe heart disease (episodes of ischemic heart disease in the last 6 months, cardiac arrhythmia or heart failure)
* Medical history of sarcoidosis or parathyroid disease
* History of malabsorption syndrome (for example pancreatic insufficiency, celiac disease or Crohn's disease), history of small bowled resection or any medical condition that may interfere with Vitamin D absorption
* Patients who are expected to administer nutritional supplements containing Vitamin D, or who are being treated with drugs (or combination of drugs) that contain Vitamin D
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Analysis of gene expression in urothelial tumor tissue, comparing initial tumor biopsy and cystectomy tumor tissue exposed to Vitamin D (reported in number of mRNA copies) | One year post-cystectomy
  Measurement of mRNA levels of differentiation and Vitamin D response markers (FGFR3, CDH1, CDKN1A/p21, THBD, VDR, G0S2 and GAPDH), determined by quantitative reverse transcription PCR (RT-qPCR)
Analysis of protein expression in urothelial tumor tissue, comparing initial tumor biopsy and cystectomy tumor tissue exposed to Vitamin D (reported in arbitrary units) | One year post-cystectomy
  Measurement of expression and distribution of differentiation and Vitamin D response markers (FGFR3, CDH1, CDH2, VDR, Ki67, CDKN1A/p21, KRT5, KRT14, KRT20 and UPK), determined by immunohistochemistry (IHC)

SECONDARY OUTCOMES:
Analysis of gene expression in peripheral blood leukocytes (reported in number of mRNA copies) | One to five months post-cystectomy
  Changes in the expression of Vitamin D target genes (CD14, CAMP, THBD and GAPDH) of peripheral leukocytes, determined by quantitative reverse transcription PCR (RT-qPCR)
Levels of serum 25(OH)Vitamin D (reported in ng/ml) | Ten weeks
  Determination of serum 25(OH)Vitamin D for pharmacokinetics study. First Vitamin D level will be obtained at screening visit and last Vitamin D level at the end of the study 4 weeks post-cystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Xavier Real, MD, PhD, Study Chair — Centro Nacional de Investigaciones Oncologicas CARLOS III (CNIO); Albert Font Pous, MD, PhD, Study Director — Institut Català Oncologia (ICO)
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain